CLINICAL TRIAL: NCT00047996
Title: Human Specimen Collection to Support Basic and Clinical Research
Brief Title: Blood Collection for Research Related to Certain Diseases Involving Blood Vessels
Status: Enrolling by invitation | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030015; 03-H-0015
Record Dates: First submitted 2006-07-11; First posted 2002-10-23 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-10-01

CONDITIONS: Sickle Cell Disease
Keywords: DNA; Endothelial Function; Leukocyte Gene Expression; RNA; Natural History; Sickle Cell; Coronary Artery Disease; CAD; Healthy Volunteer; HV
MeSH Terms: conditions — Anemia, Sickle Cell; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group1: Clinical Center Patients, Healthy Volunteers

SUMMARY:
The collection of human specimens from both patients and healthy volunteers is necessary for the development of laboratory assays to further basic and clinical research studies. This protocol defines the purposes for which specimens will be collected and establishes general conditions under which sample collection will be performed.

DETAILED DESCRIPTION:
The collection of human specimens from both patients and healthy volunteers is necessary for the development of laboratory assays to further basic and clinical research studies. This protocol defines the purposes for which specimens will be collected and establishes general conditions under which sample collection will be performed.

ELIGIBILITY:
* INCLUSION CRITERIA:

Males or females of age 18 years and older can be included in the study.

EXCLUSION CRITERIA:

Individuals without sickle cell disease or other chronic anemias who wish to donate blood will be excluded if the hemoglobin is less than 10 g/dL for women or less than 12g/dL for men.

Individuals with sickle cell disease or other chronic anemias will be excluded from donating blood samples if the hemoglobin is less than 6 g/dL.

A participant s most recent CBC result, obtained in the past 12 months, will be used to determine eligibility.

There are no exclusion criteria for participants donating urine.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal subjects, Male/Female
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2002-11-04 (Actual)

PRIMARY OUTCOMES:
evaluating the role of nitric oxide, inflammatory mediators, and endothelial function in inflammatory diseases of the vasculature such as sickle cell disease, coronary artery disease, pulmonary vascular or advanced lung disease, malaria, and sep...

CONTACTS AND LOCATIONS:
Overall Officials: Swee Lay Thein, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - INOVA Fairfax Hosptial, Fairfax, Virginia

REFERENCES:
- [Derived] Tumburu L, Ghosh-Choudhary S, Seifuddin FT, Barbu EA, Yang S, Ahmad MM, Wilkins LHW, Tunc I, Sivakumar I, Nichols JS, Dagur PK, Yang S, Almeida LEF, Quezado ZMN, Combs CA, Lindberg E, Bleck CKE, Zhu J, Shet AS, Chung JH, Pirooznia M, Thein SL. Circulating mitochondrial DNA is a proinflammatory DAMP in sickle cell disease. Blood. 2021 Jun 3;137(22):3116-3126. doi: 10.1182/blood.2020009063. PMID 33661274
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2003-H-0015.html